CLINICAL TRIAL: NCT01869231
Title: Evaluating the Efficacy of Current Treatments for Reducing Postoperative Ileus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Dott.ssa Angela Inviati, M.D., Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 17070401
Record Dates: First submitted 2013-05-27; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Post-operative Ileus
MeSH Terms: interventions — Olive Oil; Chewing Gum; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- major surgery (Experimental): colic surgery
  Interventions: Dietary Supplement: olive oil; Dietary Supplement: olive oil and chewing gum; Dietary Supplement: chewing gum; Dietary Supplement: water
- minor surgery (Experimental): appendectomy; cholecystectomy
  Interventions: Dietary Supplement: olive oil; Dietary Supplement: olive oil and chewing gum; Dietary Supplement: chewing gum; Dietary Supplement: water
- ileostomy and colostomy (Experimental): ileostomy colostomy
  Interventions: Dietary Supplement: olive oil; Dietary Supplement: olive oil and chewing gum; Dietary Supplement: chewing gum; Dietary Supplement: water
- other surgery (Experimental): all of others abdominal surgical intervention
  Interventions: Dietary Supplement: olive oil; Dietary Supplement: olive oil and chewing gum; Dietary Supplement: chewing gum; Dietary Supplement: water

INTERVENTIONS:
Dietary Supplement: olive oil
Dietary Supplement: olive oil and chewing gum
Dietary Supplement: chewing gum
Dietary Supplement: water

SUMMARY:
Aim was to investigate efficacy of current treatments - water, chewing gum, and olive oil, in resolving postoperative ileus.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent abdominal surgery for non neoplastic diseases

Exclusion Criteria:

* Metastatic disease
* History of inflammatory bowel disease
* Postoperative fever
* Gastrointestinal fistula
* Mint or olive allergy; and/or
* Earlier abdominal radiation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
time to flatus | two days

SECONDARY OUTCOMES:
time to stool | five days

OTHER OUTCOMES:
length of hospital stay | seven days

CONTACTS AND LOCATIONS:
Locations (1):
- Università di palermo, Palermo, Italy

REFERENCES:
- [Result] Matros E, Rocha F, Zinner M, Wang J, Ashley S, Breen E, Soybel D, Shoji B, Burgess A, Bleday R, Kuntz R, Whang E. Does gum chewing ameliorate postoperative ileus? Results of a prospective, randomized, placebo-controlled trial. J Am Coll Surg. 2006 May;202(5):773-8. doi: 10.1016/j.jamcollsurg.2006.02.009. PMID 16648017
- [Derived] Bonventre S, Inviati A, Di Paola V, Morreale P, Di Giovanni S, Di Carlo P, Schifano D, Frazzetta G, Gulotta G, Scerrino G. Evaluating the efficacy of current treatments for reducing postoperative ileus: a randomized clinical trial in a single center. Minerva Chir. 2014 Feb;69(1):47-55. PMID 24675245
- See also: Related Info — http://emedicine.medscape.com/article/178948-treatment